# **Study Title**

Effect of Arthroscopic Microfracture Combined with Stromal Vascular Fraction Therapy on Clinical and Radiological Outcomes in Gonarthrosis: A Prospective Randomized Controlled Trial

## **NCT Number**

NCT07112885

## **Organization**

Istanbul University, Department of Orthopedics and Traumatology

### **Document Date**

January 20, 2023 (The date on the cover page (January 20, 2023) was intentionally indicated to reflect the official ethics committee approval date of the study protocol, as required for regulatory documentation)

#### **Informed Consent Form**

Study Title: Effect of Arthroscopic Microfracture Combined with Stromal Vascular Fraction Therapy on Clinical and Radiological Outcomes in Gonarthrosis: A Prospective Randomized Controlled Trial Institution: Istanbul University, Department of Orthopedics and Traumatology

#### Introduction

You are invited to participate in a clinical study investigating the effects of stromal vascular fraction (SVF) injection with and without microfracture in patients with moderate knee osteoarthritis. Before you decide, it is important that you understand the purpose of the study, what it involves, and any possible risks or benefits.

## **Purpose of the Study**

The purpose of this study is to compare the clinical and radiological outcomes of two different treatment methods in patients with moderate knee osteoarthritis: (1) arthroscopic debridement and microfracture followed by intra-articular SVF injection, and (2) arthroscopic debridement followed by SVF injection alone.

#### **Procedures**

If you agree to participate, you will be randomly assigned to one of two groups. All patients will undergo arthroscopic knee debridement. All participants will undergo arthroscopic debridement. Group A will receive additional microfracture and SVF injection, while Group B will receive SVF injection alone. Follow-up visits will be conducted at baseline, 3, 6, 12, and 24 months, with MRI imaging performed at baseline, 12, and 24 months.

#### **Risks and Discomforts**

Possible risks include pain, swelling, stiffness, or infection after the procedure. As with any surgical or injection procedure, there is a small risk of complications related to anesthesia or the intervention itself.

#### **Benefits**

Potential benefits may include reduced pain, improved knee function, and possible improvement in cartilage quality. However, there is no guarantee of direct personal benefit.

## Confidentiality

All information collected during the study will be kept strictly confidential. Your identity will not be disclosed in any publication or report.

## **Voluntary Participation**

Participation in this study is entirely voluntary. You may refuse to participate or withdraw at any time without giving a reason, and this will not affect your standard medical care.

### **Contact Information**

If you have any questions or concerns about the study, please contact the principal investigator: Dr. Mehmet Yağız Yenigün Istanbul University, Department of Orthopedics and Traumatology

#### Consent

| I have read an | d understood the | e information إ | provided abo | ve. I voluntari | ly agree to | participate i | in this |
|---|---|---|---|---|---|---|---|
| study. | | | | | | | |

| Date: |
|-------|

### **Ethical Considerations**

The study protocol was approved by the Institutional Review Board of Istanbul University. All patients provided written informed consent prior to participation.



T.C. İSTANBUL ÜNİVERSİTESİ İstanbul Tıp Fakültesi Dekanlığı Klinik Araştırmalar Etik Kurulu



Sayı :E-29624016-050.99-1603453 Konu :Doç. Dr. Ömer Naci ERGİN hk.

> Sayın Doç. Dr. Ömer Naci ERGİN Ortopedi ve Travmatoloji Anabilim Dalı

İlgi : Ortopedi ve Travmatoloji Anabilim Dalının 06/04/2022 gün ve 839487 sayılı yazısı

Sorumlu araştırıcılığını üstlendiğiniz ve Dr. Mehmet Yağız YENIGÜN' ün yürüteceği 2023/106 dosya numaralı "Izole eklemiçi SVF(Stromal Vacular Fraction-Kök hücre) tedavisinin Artroskopik Mikrokırık (Debridman)-SVF tedavisinin klinik ve radyolojik sonuçları ile karşılaştırılması" başlıklı calışma, kurulmuzun 2001/2023 tarih ve 02 sayılı toplantısında görüşülerek etik yönden uygun bulunmuş olup, tutanaklar ekte sunulmuştur.

Bilgilerinizi rica ederim.

Prof. Dr. Ali Yağız ÜRESİN Kurul Başkanı

Bu belge, güvenli elektronik imza ile imzalanmıştı

Belge Doğrulama Kodu :BSNV6R250P Pin Kodu :42152 B Istanbul Tip Fakültesi Dekanlığı Çapa/FatihİSTANBU. Tel: 0 212 414 21 38/414 20 00-31561 Faks : 0 212 414 21 38 / 635 11 93 -posta : itf-dokanlık@istanbul.edu.tr Elektronik Ağ : http://istanbultip.istanbul.edu.tr dresi : https://www.turkiye.gov.tr/is Bilgi için : Cihan KILIÇ Dahili : 31346

Bu belge 5070 sayılı Elektronik İmza Kanununun 5. Maddesi gereğince güvenli elektronik imza ile imzalanmıştı

Reference: Letter of the Department of Orthopedics and Traumatology dated 06/04/2022 and numbered 839487

The study titled "Comparison of the Clinical and Radiological Outcomes of Isolated Intra-articular SVF (Stromal Vascular Fraction-Stem Cell) Therapy with Arthroscopic Microfracture (Debridement) + SVF Therapy", with file number 2023/106, for which you are the principal investigator and conducted by Dr. Mehmet Yağız YENİGÜN, was reviewed at the meeting of our committee dated 20/01/2023 and numbered 02, and it was found to be ethically appropriate. The minutes of the meeting are attached.

For your information.

**Document Verification Code: BSNV6R250P** 

**PIN Code: 42152** 

Prof. Dr. Ali Yağız ÜRESİN Chairman of the Committee

#### Note:

A subsequent ethics committee application was submitted in order to increase the number of participants (from 40 to 50) and to update the study title. This amendment request was reviewed and approved by the committee, confirming that both the protocol modification and the revised sample size were ethically appropriate.



T.C. İSTANBUL ÜNİVERSİTESİ İstanbul Tıp Fakültesi Dekanlığı Klinik Araştırmalar Etik Kurulu



Sayı :E-29624016-050.99-3285507 Konu :Doç. Dr. Ömer Naci ERGİN hk

Savın Doc. Dr. Ömer Naci ERGİN

İlgi : Ortopedi ve Travmatoloji Anabilim Dalının 17/03/2025 gün ve 3241799 sayılı yazısı

Sorumlu araştırıcılığını üstlendiğiniz ve Dr. Mehmet Yağız YENIGÜN' ün yürüteceği 2023/106 dosya numaralı "Izole eklemiçi SVF(Stromal Vacular Fraction-Kök hücre) tedavisinin Artroskopik Mikrokrık (Debridman)-SVF tedavisinin klinik ve radyolojik sonuçları ile karşılaştırılması" başlıklı çalışma, kurulumuzun 20/01/2023 tarih ve 02 sayılı toplantısında görüşülerek etik yönden uygun bulunmuştur.

İlgili değişiklik isteminiz, Değişiklik Bilgi Formu, Gönüllü sayısına ilişkin değişiklik, Tez isim eleğişikliği "İzole eklem içi SVF tedavisinin Artroskopik debridman + SVF tedavisinin klinik sonuçları ekarşılaştırılması" Tez qalışmasını "Gonartroz Hastalarında Stromal Vasküler Fraksiyon Tedavisinde ırtroskopik Mikrokırık ile Kombinasyonun Klinik ve Radyolojik Sonuçları: Randomize Kontrolük rospektif Çalışma" olarak değişirilmesi hakkında, kurdumuzun 18/04/2025 tarih ve 08 sayılı oplantısında yeniden görüşülerek etik yönden uygun bulunmuş olup, tutanaklar ekte sunulmuştur.

Bilgilerinizi rica ederim.

Prof. Dr. Ali Yağız ÜRESİN Kurul Başkanı

Ek:İstanbul Tıp Fakültesi Klinik Araştırmalar Etik Kurulu Karar Formu

edge Desperlation Koda 1898/BPA43K Pin Koda 26213 Belage Takip Adresi : Stope-//www. tember Tyr Faddiren Dekenligh Cope-Fatel-KETANDEL Belag için C. 6 1888 (2014) Belag i



**Reference:** Letter of the Department of Orthopedics and Traumatology dated 17/03/2025 and numbered 3241799

The study titled "Comparison of the Clinical and Radiological Outcomes of Isolated Intra-articular SVF (Stromal Vascular Fraction—Stem Cell) Therapy with Arthroscopic Microfracture (Debridement) + SVF Therapy", with file number 2023/106, for which you are the principal investigator and conducted by Dr. Mehmet Yağız YENİGÜN, was reviewed at the meeting of our committee dated 20/01/2023 and numbered 02, and was found to be ethically appropriate.

Your request for amendment, including the Amendment Information Form, the change in the number of participants (from 40 to 50), and the thesis title modification from "Comparison of the Clinical Outcomes of Isolated Intra-articular SVF Therapy with Arthroscopic Debridement + SVF Therapy" to "Effect of Arthroscopic Microfracture Combined with Stromal Vascular Fraction Therapy on Clinical and Radiological Outcomes in Gonarthrosis: A Prospective Randomized Controlled Trial", was reconsidered at the meeting of our committee dated 18/04/2025 and numbered 08, and was also found ethically appropriate. The minutes of the meeting are attached.

For your information.

**Document Verification Code: BS93BP48J8C** 

**PIN Code: 26213** 

Prof. Dr. Ali Yağız ÜRESİN Chairman of the Committee